CLINICAL TRIAL: NCT01593397
Title: Adiponectin Polymorphisms, Insulin Resistance, and Pharmacokinetics in Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Jerry Ingrande, Instructor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1K23GM100273-01 (NIH); 5K23GM100273-04 (NIH)
Record Dates: First submitted 2012-04-30; First posted 2012-05-08 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Obesity
Keywords: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propofol and Fentanyl administration (Experimental): Propofol and Fentanyl will be administered to all subjects. All subjects will have blood drawn to determine pharmacokinetic variables. Processed EEG will be used to determine pharmacodynamics. Plasma samples will be used to ascertain adiponectin levels and for DNA sampling for analysis of adiponectin single nucleotide polymorphisms.
  Interventions: Drug: Propofol and Fentanyl administration

INTERVENTIONS:
Drug: Propofol and Fentanyl administration — Propofol will be administered to all patients via infusion at a dose of 2 mg/kg lean body weight/minute. The infusion will stop once loss of consciousness is reached. Fentanyl will be administered via target controlled infusion to achieve a plasma concentration of 2 ng/ml.
  Other Names: anesthetic administration

SUMMARY:
The primary objective of this study is to determine the influence of insulin resistance on drug metabolism and response in obese subjects. The investigators hypothesize that expression of adiponectin (a hormone secreted by fat tissue), and specific variants in the adiponectin gene can predict the insulin resistance and drug response among obese subjects.

DETAILED DESCRIPTION:
The following study will hypothesizes that insulin resistance causes changes in drug metabolism, elimination, and effect. We will differentiate the insulin resistant phenotype amongst obese individuals on the basis of both laboratory (fasting insulin, triglycerides, fasting glucose) analysis, and quantitative and qualitative adiponectin expression. We will determine the effect of insulin resistance on the pharmacokinetics and pharmacodynamics of anesthetic induction agents and opioids, using propofol and fentanyl as examples.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include patients of adult age
* American Society of Anesthesiologists Class I, II, or III, and undergoing elective surgical procedures requiring general anesthesia
* Body mass index greater than 35

Exclusion Criteria:

* Patients with evidence of hepatic, renal, or cardiovascular dysfunction
* History of difficult tracheal intubation, or adverse reaction to anesthesia shall be excluded from the study
* Patients taking prescribed or over-the-counter anxiolytics, narcotics, or sleeping aids, will also be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
plasma concentration of drugs fentanyl and propofol | measured for 12 hours (beginning of anesthesia to 12 hours after)
  Plasma concentration over time will be measured and modeled in order to calculate drug clearance, volume of distribution, area under the curve, and micro rate constants.
  Knowledge of these variables will allow safer administration of anesthetic drug administration in the obese population.

SECONDARY OUTCOMES:
Adiponectin plasma protein levels | measured once (immediately before the operation)
  The investigators will measure specific levels of the protein adiponectin in the blood, to determine if quantitative expression of adiponectin can predict insulin resistance in obesity and drug metabolism and response.
Adiponectin gene polymorphisms | measured once per study (immediately before the operation)
  The investigators will look at specific genetic variants of the adiponectin gene to determine if expression of specific variants can predict insulin resistance and changed in drug response and metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Ingrande, M.D., M.S., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Department of Anesthesia, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
pharmacokinetic models will be published after data analysis and study completion